CLINICAL TRIAL: NCT04545632
Title: A Multi-center, Prospective, Observational Study to Evaluate Ethanol-induced Symptoms in Patients With Chemotherapy of Docetaxel
Brief Title: Docetaxel Ethanol-induced Symptoms; The Incidence and Risk Forecating Factor
Acronym: DETECT
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-DTX-OS-401
Record Dates: First submitted 2020-07-08; First posted 2020-09-11 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; NSCLC; Prostate Cancer; Head and Neck Cancer; Gastric Cancer; Esophageal Cancer; Ovarian Cancer
Keywords: Chemotherapy; Ethanol-containing docetaxel
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients receiving chemotherapy with ethanol-containing docetaxel

SUMMARY:
To determine the incidence and risk factors of ethanol-induced symptoms, this multicenter, prospective, observational study is designed to include patients in Korea who are receiving chemotherapy with ethanol-containing docetaxel alone or in combination. Subjects who voluntarily provide written informed consent to provide information for this study and meet the inclusion/exclusion criteria will be given an enrollment number and will be followed during the observation period to collect study-related data in the Case Report Forms (CRFs) as predefined in the study protocol. Patients' decision to participate (or not) in this study will not affect their treatment (physician's prescriptions or diagnostic/therapeutic decisions).

DETAILED DESCRIPTION:
Ethanol-induced symptoms questionnaire will be administered three times during the baseline visit (Visit 1) - before, during, and within 30 minutes after treatment with docetaxel - and then during the follow-up visit (or phone call) at 24 hours after the treatment. There will be no restrictions as to what concomitant medications can be used before and after treatment with ethanol-containing docetaxel, and investigators will determine the manufacturer, preparation method, and dosage regimen of docetaxel as per routine care at their study site.

The following data will be collected:

* Demographics (gender, age, drinking history)
* Height, body weight and body mass index (BMI)
* Cancer-related data (diagnosis, date of diagnosis)
* ECOG PS
* Underlying diseases
* Prior and concomitant medications
* Data on docetaxel therapy (timing of initiation of the chemotherapy, monotherapy/combination therapy, intervals between chemotherapy treatments, product name, dose (mg), administered ethanol dose (g), blood alcohol content (BAC*), type and volume of intravenous (IV) fluid administered before and after treatment and fluid mixed with docetaxel, duration of injection)

  * Blood alcohol content (BAC): Widmark formula = administered ethanol dose (g) / body weight (kg) × gender constant (0.68 for males and 0.55 for females)
* Ethanol-induced symptoms questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide written informed consent to collect and use personal information after an explanation of the objectives and methods of the study
2. Adult males and females aged 19 years and older
3. Chemotherapy with ethanol-containing docetaxel (≥50 mg/m2) alone or in combination for a pathologically confirmed cancer
4. ECOG Performance Status (ECOG PS) scores ≤2
5. Patients who are capable of understanding the questionnaire items and directly answering questions

Exclusion Criteria:

1. History of psychiatric disorder, seizure, or central nervous system disorder
2. Metastasis to the central nervous system (although patients without neurological symptoms are eligible)
3. Active hepatitis
4. Individuals who meet any of the following:

   * AST/ALT ≥2 X upper limit of normal (ULN)
   * Total bilirubin ≥2 X ULN
   * Hemoglobin <9.0 g/dL
5. Combination chemotherapy with ethanol-containing anticancer drugs other than docetaxel
6. Alcohol, hypnotic or tranquilizer intake within 24 hours before treatment with docetaxel
7. Pregnant or nursing women or women of childbearing potential
8. Subjects who are currently participating in another clinical trial (of drugs or medical devices) or plan to do so during the study. However, subjects are allowed to participate in another non-interventional observational study or registry study.
9. Patients who are otherwise considered by the investigator to be ineligible for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy with ethanol-containing docetaxel
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence of ethanol-induced symptoms as a whole | Time Frame : From the time of treatment started until the end of follow-up(24hours after the treatment)
  An increase from baseline in the number of ethanol-induced symptoms during or after treatment

SECONDARY OUTCOMES:
Incidence of each ethanol-induced symptom | Baseline visit - before, during, and within 30 minutes after treatment, Follow-up visit - 24 hours after the treatment
  Any increase from baseline in the number of each ethanol-induced symptom during or after treatment
Incidence of ethanol-induced symptoms as a whole during and at each time point after treatment | Baseline visit - during, and within 30 minutes after treatment, Follow-up visit - 24 hours after the treatment
  The incidence of ethanol-induced symptoms as a whole will be calculated at each post-dose time point (during, within 30 minutes after treatment, and 24 hours after treatment) compared with baseline values
Incidence of each ethanol-induced symptom during and at each time point after treatment | Baseline visit - during, and within 30 minutes after treatment, Follow-up visit - 24 hours after the treatment
  The incidence of ethanol-induced symptoms as each will be calculated at each post-dose time point (during, within 30 minutes after treatment, and 24 hours after treatment) compared with baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Myung Sook Hong, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Hanyang University Guri Hospital, Guri-si, South Korea